CLINICAL TRIAL: NCT06687915
Title: The Comparison of Balance and Coordination Between Visually Impaired and Healthy Sedentary Individuals
Brief Title: Comparison of Balance and Coordination Parameters of Visually Impaired and Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Asst. Prof., Bahçeşehir University
Other Study IDs: Study0007
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Blindness Congenital
Keywords: Complete Blindness; Visual Impairments; Posture Balance
MeSH Terms: conditions — Blindness; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Congenitally blind: Individuals with congenital visual impairment were included in this group.
- Healthy: Healthy sedentary individuals were included in this group.

SUMMARY:
The aim of this [observational study] is to examine balance in multiple aspects by comparing balance, coordination, and gait parameters between congenitally blind individuals and healthy individuals with multiple scales.

The main questions it aims to answer are:

Is there a difference in balance and coordination between congenitally blind individuals and healthy individuals? comparison group: Healthy sedated individuals Participants will be asked to complete balance scales.

DETAILED DESCRIPTION:
Visually impaired, with all corrections, individuals who have one tenth of the usual visual acuity of the seeing eye, i.e. 20/200 visual acuity or less, or whose visual angle does not exceed 20 degrees are called blind. The meaning of 20/200 is that an individual affected by visual impairment can see from 60 cm, while an individual with normal vision can see from 6 m. Narrow angle of vision means that, despite normal visual acuity, vision is limited only to the centre, 20 degrees, and objects beyond 20 degrees cannot be seen.

Balance depends on the integration of information received from proprioceptive, vestibular and visual sensory systems. It has been observed that visually impaired individuals have problems in postural stability and balance due to insufficient information from the visual system. In this study, it was aimed to compare the balance, coordination and gait parameters of congenitally visually impaired individuals and healthy sedentary individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Congenital visual impairment
* Not having any acute or chronic disease other than congenital blindness

Exclusion Criteria:

* Having musculoskeletal deformity
* Being involved in a professional sport
* Having received physiotherapy treatment for balance before

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this study, congenitally visually impaired individuals and healthy individuals aged between 18-40 years were included.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Test | At the baseline of the study
  Berg Balance Scale was developed for postural control assessment. It includes 14 instructions and for each instruction, the patient's performance is observed and a score between 0-4 is given. It takes between 10 and 20 minutes to complete the scale

CONTACTS AND LOCATIONS:
Overall Officials: Emine Atıcı, Assoc. Prof., Study Director — Okan University; Alper Percin, Ph.D., Principal Investigator — Bahçeşehir University
Locations (1):
- Avrasya University, Trabzon, Ortahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It can be shared at the request of the researchers.

REFERENCES:
- [Background] Blum L, Korner-Bitensky N. Usefulness of the Berg Balance Scale in stroke rehabilitation: a systematic review. Phys Ther. 2008 May;88(5):559-66. doi: 10.2522/ptj.20070205. Epub 2008 Feb 21. PMID 18292215
- [Background] Chen EW, Fu AS, Chan KM, Tsang WW. The effects of Tai Chi on the balance control of elderly persons with visual impairment: a randomised clinical trial. Age Ageing. 2012 Mar;41(2):254-9. doi: 10.1093/ageing/afr146. Epub 2011 Dec 16. PMID 22180415
- [Background] Gleeson M, Sherrington C, Lo S, Keay L. Can the Alexander Technique improve balance and mobility in older adults with visual impairments? A randomized controlled trial. Clin Rehabil. 2015 Mar;29(3):244-60. doi: 10.1177/0269215514542636. Epub 2014 Jul 15. PMID 25027444